CLINICAL TRIAL: NCT00135538
Title: Does Chronic Ventilatory Support Improve the Outcomes of Rehabilitation in Hypercapnic COPD Patients?
Brief Title: The Additional Value of Noninvasive Ventilation Next to Rehabilitation in Hypercapnic COPD Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groningen Research Institute for Asthma and COPD (Other)
Collaborators: The Netherlands Asthma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECOVER1
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Intermittent Positive-Pressure Ventilation; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Noninvasive positive pressure ventilation

SUMMARY:
The purpose of this study is to investigate whether noninvasive ventilation by nose mask during the night has additional benefits next to pulmonary rehabilitation in patients with severe hypercapnic COPD.

DETAILED DESCRIPTION:
Several randomised controlled trials in patients with stable Chronic Obstructive Pulmonary Disease (COPD) have demonstrated that pulmonary rehabilitation (PR) improves dyspnoea, exercise tolerance, and health-related quality of life. Research in this field has been important in our department for several years. The first study in this respect was started in 1986 comparing outpatient rehabilitation with rehabilitation in the community in patients with severe COPD. This study showed that rehabilitation supervised by a physical therapist in the community is effective for a long period in contrast to outpatient rehabilitation. In 1990 the second study started showing that positive initial benefits of home based rehabilitation on quality of life can be maintained for 18 months if the patients visit the local physical therapist once a month.

However, less positive effects of rehabilitation have been reported in the more severe patients. Because of dyspnoea due to inspiratory muscle fatigue patients may not receive an adequate training stimulus, and therefore rehabilitation might be less effective. In these more severe patients alternative therapies are needed. These non-pharmacological treatments include nutritional supplementation, oxygen therapy, lung transplantation, lung volume reduction surgery and ventilatory support.

The last few years a discussion within the 4 home mechanical ventilation centres (HMV) in the Netherlands has been started about the role of chronic ventilatory support in end-stage COPD. Theoretically, it might be effective because:

1. a resetting of the respiratory centre may reduce daytime PaCO2;
2. a better internal milieu (pH, PaO2, PaCO2) may improve peripheral muscle function;
3. resting the respiratory muscles during the night may increase their daytime strength and endurance;
4. a reduction in the number of nocturnal arousals may improve the quality of sleep. Nevertheless, none of these mechanisms has been proven and currently there is no evidence that noninvasive positive pressure ventilation (NIPPV) should be given to stable patients with COPD. While several randomised controlled trials (RCT's) on NIPPV have been published with different outcomes, a recent meta-analysis did not show beneficial effects on blood gasses, lung function, respiratory muscle function and walking distance.

In contrast several uncontrolled studies did show clear benefits from NIPPV on gas-exchange, dyspnoea and quality of life. Possible reasons for these conflicting outcomes are differences in:

1. selection of patients,
2. adequacy of ventilatory support,
3. length of ventilatory support. Interestingly, it seems that studies with a positive outcome included mainly patients with hypercapnia, suggesting this as an important selection criterion.

The hypothesis is that long term NIPPV in hypercapnic patients with COPD may improve the effects of rehabilitation at home regarding health status, ADL function, dyspnoea and exercise tolerance. Secondly, we like to elucidate the exact mechanisms why NIPPV might be effective in this group of patients.

Comparison: patients who receive noninvasive ventilation during the night while following a pulmonary rehabilitation program with patients who only follow a rehabilitation program without receiving the noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1< 50%, Tiffeneau < 70%)
* Dyspnoea on exertion and a reduced exercise capacity
* Age 75 years or less
* PaCO2 > 6.0 kPa at rest without oxygen

Exclusion Criteria:

* Cardial/neuromuscular diseases limiting a successful rehabilitation
* Obstructive sleep apnoea syndrome: apnea/hypopnea index (AHI) > 10
* Previous exposure to chronic NIPPV
* Participation in a pulmonary rehabilitation program less than 18 months ago

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-11; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life measured by the Chronic Respiratory Questionnaire

SECONDARY OUTCOMES:
Activities of daily Living
Dyspnea (Medical Research Council Scale [MRC], baseline dyspnea index [BDI], Borg)
Exercise tolerance (Cycle ergometer test, 6-minute walk distance [6-MWD], incremental shuttle walking test [ISWT], endurance shuttle walking test [ESWT])
Pulmonary function testing
Sleep quality (polysomnography)
Respiratory muscle activity (endurance shuttle walking test [EMG])
Respiratory muscle strength (PImax, PEmax)

CONTACTS AND LOCATIONS:
Overall Officials: Marieke L Duiverman, Principal Investigator — University Medical Center Groningen
Locations (1):
- University medical Hospital Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Altenburg WA, Duiverman ML, Ten Hacken NH, Kerstjens HA, de Greef MH, Wijkstra PJ, Wempe JB. Changes in the endurance shuttle walk test in COPD patients with chronic respiratory failure after pulmonary rehabilitation: the minimal important difference obtained with anchor- and distribution-based method. Respir Res. 2015 Feb 19;16(1):27. doi: 10.1186/s12931-015-0182-x. PMID 25849109
- [Derived] Duiverman ML, Wempe JB, Bladder G, Vonk JM, Zijlstra JG, Kerstjens HA, Wijkstra PJ. Two-year home-based nocturnal noninvasive ventilation added to rehabilitation in chronic obstructive pulmonary disease patients: a randomized controlled trial. Respir Res. 2011 Aug 23;12(1):112. doi: 10.1186/1465-9921-12-112. PMID 21861914
- [Derived] Duiverman ML, Wempe JB, Bladder G, Jansen DF, Kerstjens HA, Zijlstra JG, Wijkstra PJ. Nocturnal non-invasive ventilation in addition to rehabilitation in hypercapnic patients with COPD. Thorax. 2008 Dec;63(12):1052-7. doi: 10.1136/thx.2008.099044. Epub 2008 Aug 18. PMID 18710905
- [Derived] Duiverman ML, Wempe JB, Bladder G, Kerstjens HA, Wijkstra PJ. Health-related quality of life in COPD patients with chronic respiratory failure. Eur Respir J. 2008 Aug;32(2):379-86. doi: 10.1183/09031936.00163607. Epub 2008 Apr 2. PMID 18385168